CLINICAL TRIAL: NCT02435667
Title: Resistance Exercise Training in Heart Failure With Preserved Ejection Fraction (Resist - HFpEF)
Brief Title: Resistance Training in HFpEF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Thomas P. Olson, M.S., Ph.D., Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 15-000320
Record Dates: First submitted 2015-04-29; First posted 2015-05-06 (Estimated); Last update posted 2021-02-03 (Actual); Status verified 2021-02

CONDITIONS: Heart Failure Preserved Ejection Fraction
Keywords: Resistance Training; Exercise; Heart Failure preserved Ejection Fraction
MeSH Terms: conditions — Heart Failure, Diastolic; Motor Activity | interventions — Resistance Training; Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Resistance Exercise Training (Experimental): Entails 36 supervised resistance exercise training sessions (3 sessions per week for 12 weeks). Each exercise session will be supervised by a trained, certified Exercise Physiologist specializing in Cardiac Rehabilitation. The specific resistance exercise training will include Aerobic Exercise, Resistance Exercise, and Core Strengthening Exercises. Other baseline and follow-up tests include: DEXA bone scan, Blood Draw, Cardiopulmonary Max Exercise Test, Quality of Life Questionnaire, and a Submaximal Exercise Test.
  Interventions: Other: Resistance Exercise Training; Radiation: DEXA bone scan; Other: Cardiopulmonary Max Exercise Test; Other: Quality of Life Questionnaire; Other: Submaximal Exercise Test; Other: Blood Draw
- Standard Care (Placebo Comparator): No resistance exercise training. Patients will stay on their current healthcare regimen as previously assigned by their physician. Patients will still undergo baseline and follow-up tests similar to the Resistance Exercise Training group, including: DEXA bone scan, Blood Draw, Cardiopulmonary Max Exercise Test, Quality of Life Questionnaire, and a Submaximal Exercise Test.
  Interventions: Radiation: DEXA bone scan; Other: Cardiopulmonary Max Exercise Test; Other: Quality of Life Questionnaire; Other: Submaximal Exercise Test; Other: Blood Draw

INTERVENTIONS:
Other: Resistance Exercise Training — 1. Aerobic Exercise
     a. Each participant will engage in 5 minutes of aerobic based exercise on an arm/leg ergometer (NuStep Cross Trainer) at an intensity of 12-14 on the Borg Rating of Perceived Exertion Scale as a warm-up prior to the exercise session and again as a cool-down at the end of the exercise session.
  2. Resistance Exercise - 2 sets of 8-12 repetitions - beginning at 60% of the initial 1 RM.
     a) Leg Extension, b) Bicep Curl, c) Leg Press, d) Chest Press, e) Leg Curl, f)Seated Row (horizontal or pulldown), g) Calf Raises
  3. Core Strengthening Exercises a. 5-10 minutes of stability ball and balance exercises
  Arms: Resistance Exercise Training
Radiation: DEXA bone scan — A DEXA scan that provides bone density measures.
Other: Cardiopulmonary Max Exercise Test — Pedaling on a cycle ergometer to volitional fatigue.
Other: Quality of Life Questionnaire — A 10 minute questionnaire that measures quality of life.
Other: Submaximal Exercise Test — Two short submaximal constant-load exercise sessions at 20 Watts. Each session will include 6 minutes of cycling (baseline). Following baseline, the sessions will be randomized to continued constant-load cycling for an additional 9 minutes (for echocardiographic measures) or randomized sub-systolic inflation of bilateral thigh pressure tourniquets to 40 and 80 mmHg for 3 minutes with 3 minutes of deflation between inflations to stimulate locomotor muscle neural feedback.
Other: Blood Draw — A blood draw amounting to 1 teaspoon of blood drawn.

SUMMARY:
The objective of this proposal is to determine the effect of resistance exercise training on locomotor muscle function, exercise capacity, exertional symptoms, and quality of life in HF patients with preserved ejection fraction (HFpEF).

DETAILED DESCRIPTION:
In this randomized controlled pilot study of resistance exercise training in patients with HFpEF, the investigators will recruit 24 HFpEF patients who will be randomized to resistance exercise training (RT - n=12) or no resistance exercise training (standard care control group [CTL] - n=12). The investigators will have baseline and follow-up measures of clinical characteristics, leg muscle strength, quality of life, lean muscle mass (body composition via DXA including segmental lean mass), maximal cardiopulmonary exercise test (peak VO2, peak work, ventilatory efficiency), constant-load submaximal cardiopulmonary exercise test with speckle tracking echocardiography (exertional dyspnea and fatigue at matched workloads, cardiac output, diastolic function, left ventricular strain, ventilation, gas exchange, and locomotor muscle neural feedback).

Participants will be asked to make 4 separate study visits. Those randomized to undergo Resistance Training will be expected to make those visits as well.

ELIGIBILITY:
All patients will be managed by their primary care physician or cardiologist with additional review and oversight by Dr. Borlaug (Co-Investigator) prior to enrollment to ensure adequacy of inclusion and exclusion criteria and that participation in exercise testing and resistance exercise training is safe.

Inclusion Criteria, includes:

* Clinical diagnosis of HFpEF.
* Patients 18-80 yrs old with a history stable (no medication changes in past 6 weeks (w/duration of diagnosis >6 months).
* New York Heart Association class I-III.
* Ejection fraction ≥40%.
* Current non-smokers with <15 pack year history.
* Non-pregnant women, and individuals who are able to exercise (i.e. without orthopedic limitations or neuromuscular disorders).

Exclusion Criteria, includes:

* Patient refusal to participate.
* Significant orthopedic or neuromuscular limitations
* Significant cognitive impairment
* Hemoglobin < 7.0 g/d.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2015-06 (Actual); Primary Completion 2021-01 (Actual); Study Completion 2021-01 (Actual)

PRIMARY OUTCOMES:
Bone density and strength | 12 weeks
  DEXA scan
Cardiopulmonary Function | 12 weeks
  Cardiopulmonary bike exercise
Quality of Life | 12 weeks
  Questionnaire
Blood Biomarkers | 12 weeks
  Blood draw

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Olson, MS, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials